CLINICAL TRIAL: NCT07055854
Title: Virtual Mindful After Cancer Intervention to Promote Sexual Health for Breast and Gynecologic Cancer Survivors
Brief Title: Virtual Mindful After Cancer (MAC) Intervention to Promote Sexual Health for Breast and Gynecologic Cancer Survivors
Acronym: MAC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jessica Gorman, Associate Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HE-2023-492; 1R34CA286710 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-07-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gynecologic Cancers; Breast Cancer
Keywords: cancer survivorship; mindfulness; sexual health; intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Mindful After Cancer Program

INTERVENTIONS:
Behavioral: Mindful After Cancer Program — The Mindful After Cancer Program provides education, mindfulness training, and peer support to help cancer survivors navigate sexual and body image concerns.
  Arms: Intervention

SUMMARY:
The goal of this study is to plan for a large scale evaluation of a program called Mindful After Cancer, or MAC. The MAC Program provides training in mindfulness, educational material about sexual health after cancer, and support to cancer survivors experiencing sexual and body image concerns.

The main study aims are to:

1. Develop effective plans for recruiting participants across multiple sites
2. Evaluate participation in the program and surveys
3. Develop plans to train and supervise the professionals who will deliver the program.

Researchers will compare study recruitment across three sites, aiming to identify the most efficient approach for a larger future trial.

Participants who are randomly assigned to receive the MAC program will receive access to the 8-week program delivered by a trained mindfulness coach using videoconference and online materials. They will asked to participate in an interview about their experiences at the end of the program.

Participants who are not randomly assigned to the MAC program will receive access to the program's educational materials after completing the final survey.

All study participants will be asked to complete 3 online surveys. Participants randomly assigned to the MAC Program will also be asked to complete a one-on-one interview about their experience in the program.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with female breast or gynecologic cancer at stage I-IV
* Diagnosed at least 6 months ago
* At least one sexual concern in a validated screener
* Access to high speed internet via smart phone, tablet, and/or computer

Exclusion Criteria:

• Those who do not comprehend English since the MAC program is only available in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment Accrual Rate- The percent of eligible candidates who enroll | Baseline
Intervention Fidelity- The percent of required topics covered during intervention sessions as measured by completion of a checklist. | Up to 1 week post-intervention.
  Adherence to the manual is assessed by independent review of audio-recorded intervention sessions using a checklist of material to be covered in each session.
Retention Rate - The percent of enrolled participants who complete all study surveys | Up to the 3 month post-intervention survey at week 22.

SECONDARY OUTCOMES:
MAC intervention Drop Out- As measured by session attendance. | Up to completion of the 8-week MAC intervention.
  Percentage of enrolled participants who stop attending the MAC intervention arm after attending the first session.

OTHER OUTCOMES:
Exploratory outcome: Interest in sexual activity as measured by the interest in sexual activity domain from the PROMIS Sexual Function and Satisfaction Scale. | Up to the 3 month post-intervention survey at week 22.
  To compare sexual interest longitudinally after enrollment between those receiving MAC and those receiving usual care. The sexual interest domain has 2 items, Range 2-10. Higher score indicates more interest in sexual activity.
Exploratory Outcome: Body Appreciation as measured by the Body Appreciation Scale. | Up to the 3 month post-intervention survey at week 22.
  To compare body appreciation longitudinally after enrollment between those receiving MAC and those receiving usual care. The Body Appreciation Scale has13 items, Range 13-65. Higher score indicates more positive body appreciation.
Exploratory Outcome: Sexual Satisfaction as measured by the Global Measure of Sexual Satisfaction scale (GMSEX). | Up to the 3 month post-intervention survey at week 22.
  To compare sexual satisfaction longitudinally after enrollment between those receiving MAC and those receiving usual care. The GMSEX scale has 5 items, Range 5-35. Higher score indicates higher level of sexual satisfaction.
Exploratory outcome: Self-Efficacy as measured by the Self-Efficacy for Managing Chronic Disease Scale (adapted). | Up to the 3 month post-intervention survey at week 22.
  To compare self-efficacy for managing sexual health in chronic disease longitudinally after enrollment between those receiving MAC and those receiving usual care. The adapted self-efficacy for managing chronic disease scale has 6 items, Range 6-60. Higher score indicates better self-efficacy for managing sexual health after cancer.
Exploratory outcome: Self-compassion as measured by the Self-Compassion Scale Short Form (SCS-SF). | Up to the 3 month post-intervention survey at week 22.
  To compare self-compassion longitudinally after enrollment between those receiving MAC and those receiving usual care. The SCS-SF has 12 items, Range 12-60. Higher score indicates greater self-compassion for managing chronic disease scale has 6 items, Range 6-60. Higher score indicates better self-efficacy for managing sexual health after cancer.
Exploratory outcome: Mindfulness as measured by the Five-Facet Mindfulness Questionnaire (FFMQ-15). | Up to the 3 month post-intervention survey at week 22.
  To compare mindfulness longitudinally after enrollment between those receiving MAC and those receiving usual care. The FFMQ-15 has 15 items with 5 sub-scales: Observe, Describe; Act with Awareness; Non-Judgement, Non-Reactivity. Sub-scale score range 3-15. Higher score indicates greater mindfulness.
Exploratory outcome: Social support as measured by the modified Medical Outcomes Study Social Support Survey (mMOS-SS). | Up to the 3 month post-intervention survey at week 22.
  To compare social support longitudinally after enrollment between those receiving MAC and those receiving usual care. The mMOS-SS has 8 items, Range 1-5. The score for mMOS-SS is calculated as the average score of subscale items transformed to a zero to 100 scale, with higher scores indicating more support.
Exploratory outcome: Depressive Symptoms as measured by the Patient Health Questionnaire (PHQ-8) | Up to the 3 month post-intervention survey at week 22.
  To compare depressive symptoms longitudinally after enrollment between those receiving MAC and those receiving usual care. The PHQ-8 has 8 items, Range 0-24. Higher scores indicate higher levels of depressive symptoms.
Exploratory outcome: Anxiety as measured by the PROMIS Emotional Distress Anxiety Short Form 6a. | Up to the 3 month post-intervention survey at week 22.
  To compare anxiety longitudinally after enrollment between those receiving MAC and those receiving usual care. The PROMIS Emotional Distress Anxiety Short Form 6a has 6 items, Range 6-30. Higher scores indicate higher levels of anxiety.
Exploratory outcome: Quality of life as measured by the PROMIS Global Health 10. | Up to the 3 month post-intervention survey at week 22.
  To compare quality of life longitudinally after enrollment between those receiving MAC and those receiving usual care. The PROMIS Global Health 10 has 10 items, Range 10-50. Higher scores indicate better functioning.
Exploratory outcome: Sexual function (Lubrication) as measured by the lubrication domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare vaginal lubrication longitudinally after enrollment between those receiving MAC and those receiving usual care. The vaginal lubrication domain has 3 items, Range 3-15. Higher score indicates more vaginal lubrication.
Exploratory outcome: Sexual function (Vaginal Discomfort) as measured by the vaginal discomfort domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare vaginal discomfort longitudinally after enrollment between those receiving MAC and those receiving usual care. The vaginal discomfort domain has 2 items, Range 2-10. Higher score indicates more vaginal discomfort.
Exploratory outcome: Sexual function (Labia Discomfort) as measured by the labia discomfort domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare labia discomfort longitudinally after enrollment between those receiving MAC and those receiving usual care. The labia discomfort domain has 2 items, Range 2-10. Higher score indicates more labia discomfort.
Exploratory outcome: Sexual function (Clitoral Discomfort) as measured by the clitoral discomfort domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare clitoral discomfort longitudinally after enrollment between those receiving MAC and those receiving usual care. The clitoral discomfort domain has 2 items, Range 2-10. Higher score indicates more clitoral discomfort.
Exploratory outcome: Sexual function (Orgasm ability) as measured by the orgasm ability domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare orgasm ability longitudinally after enrollment between those receiving MAC and those receiving usual care. The orgasm ability domain has 1 item, Range 1-5. Higher score indicates more orgasm ability.
Exploratory outcome: Sexual function (Orgasm pleasure) as measured by the orgasm pleasure domain from the PROMIS Sexual Function and Satisfaction Scale. | From Baseline up to the 3 month post-intervention survey at week 22.
  To compare orgasm pleasure longitudinally after enrollment between those receiving MAC and those receiving usual care. The orgasm pleasure domain has 2 items, Range 2-10. Higher score indicates more orgasm pleasure.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Samaritan Pastega Regional Cancer Center, Corvallis, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No